CLINICAL TRIAL: NCT02865252
Title: The Effect of Mobilization With Movement on Pain and Function Among Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-2014-04-323
Record Dates: First submitted 2016-08-08; First posted 2016-08-12 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Osteoarthritis
Keywords: manual therapy; mobilization with movement
MeSH Terms: conditions — Osteoarthritis | interventions — Movement; Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MWM treatment (Active Comparator): Mobilization with movement (MWM) is a combination of sustained passive accessory joint mobilization with an active or functional movement.
  MWM will be applied (three sets of 10 repetitions) during active knee flexion and extension range of motion (ROM). The therapist initially will apply the pain-free manual glide force on the tibia with the knee resting in a mid-range position. The glide force will be sustained while the patient performed 10 repetitions of self-active full range knee flexion and extension; overpressure was included at the end range.
  Interventions: Other: MWM Treatment
- MWM sham (Sham Comparator): The patients will be handled similarly to MWM treatment group, except that they will not receive directional glide; instead, the physiotherapist's hands are just touch the knee skin without pressure; one hand on the tibia while the other hand on the femur. However, available active knee flexion and extension ROM will be performed (three sets of 10 repetitions).
  Interventions: Other: MWM Sham

INTERVENTIONS:
Other: MWM Treatment
  Other Names: Mobilization with Movement, Manual therapy
  Arms: MWM treatment
Other: MWM Sham
  Arms: MWM sham

SUMMARY:
Osteoarthritis (OA) is the most prevalent form of arthritis and is reported to be the most important reason behind functional disability and musculoskeletal disorders among aged individuals. OA is "a total joint failure; represented by pathological damage to articular cartilage, that affects bone, menisci, synovium, ligaments, and neuromuscular tissue". Knee OA could be responsible for pain and functional disability in 19.2% of individuals aged more than 45 years in the Framingham study and in 27.8% of such individuals in the Johnston County Osteoarthritis Project. However, in the third National Health and Nutrition Examination Survey (NHANES III), nearly 37% of individuals aged 60 years or older had radiographic knee OA. Oliveria et al. (1995) reported that age- and sex-standardized incidence rates of symptomatic hip, knee, and hand OA were 88, 240, and 100/100,000 person-years, respectively. In addition, the incidence rates of symptomatic OA of the knee, hand, or hip increased rapidly at age 50 and then levelled off beyond age 70. There were not enough data to report the prevalence of OA in Arabic countries. However, a cross-sectional study performed in Saudi Arabia demonstrated radiographic knee OA in 53.3% of men and 60.9% of women, while about 18% of women and 10% of men had symptomatic OA. Although it is well established that OA is mainly caused by damage occurring in the joint because of degeneration and inflammation, there is no known cure for OA and our understanding of the pathological aetiology of OA is still deficient and poorly understood.

The primary objective of this study is to investigate the immediate and the carry-over effect of MWM on pain and function in patients with knee OA. A secondary objective is to evaluate this effect among those patients who demonstrate features of central sensitization.

DETAILED DESCRIPTION:
Participants:

A power analysis was performed using G*Power 3.1 (F tests, analysis of variance [ANOVA]: repeated measure, within-between interaction, and a priori: compute required sample size). A result of 16 patients (treatment group = 8 and sham group = 8) was used to calculate an effect size (ES) of 0.27 for the pressure pain threshold of the knee after the intervention between groups. The power estimated for ANOVA for the two groups with a significance of 0.05 revealed that a total sample size of 27 patients was necessary to obtain a power of 0.80. Considering a 20% attrition rate, a minimum of 18 patients needed to be recruited for the first phase in this study.

Patients with knee OA who attended King Fahd Hospital of the University will be recruited for this study. Patients will be diagnosed at the orthopedic clinic and referred to the Department of Physiotherapy. Patients who are willing to participate in the study will be screened for their eligibility

Ethical considerations:

The study was approved by the Institutional Review Board (IRB) at the University of Dammam (IRB Number: IRB-2014-04-323). Eligible individuals for this study will be informed of the risks and benefits and will be asked to read and sign a written consent form.

Participant confidentiality will be maintained by using a code instead of the participant's name on the data collection form. All data collection forms will be saved in a file and secured in a locker. Only the researcher and the supervisor had a key to open this locker.

Statistical Analysis:

Data will be analyzed using International Business Machines (IBM) Statistical Package for Social Sciences (SPSS) for windows (version 20.0), significance level was set at p < 0.05.

In phase 1, patients characteristics between groups at baseline will be analyzed using an independent t-test. One way ANOVA with repeated measures will be used to analyze the differences for other parametric data, Bonferroni adjustment will be used to compare main effects. Post-hoc tests will be performed to reveal differences of within- between groups over time (baseline, immediately post intervention, and after 2 days of intervention). For Likert-scale WOMAC, the Mann-Whitney U test will be used to investigate between-group analysis. Whereas, the Wilcoxon test will be used for within-group analysis. Further analysis to reveal correlations between the outcome measures will be investigated using Pearson Correlation test.

In phase 2, the groups are matched in age, gender, and BMI. The related t-test will be used to investigate differences between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Had unilateral or bilateral knee OA
* Knee OA K&L grade ≥ 2
* VAS = 3 cm over the previous 24 hours
* Able to walk ≥ 6-meter distances with or without an aid

Exclusion Criteria:

* Had knee or lower limb surgery
* Oral corticosteroid use (current\ 4 weeks)
* Altered sensation around knee and shoulder
* Exhibited cognitive difficulties
* Intra-articular corticosteroid or hyaluronic acid injection within 6 months
* Had leg sciatica
* Contraindication to manual therapy

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-10; Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The Visual Analog Scale (VAS) | Change from Baseline in Visual Analog Scale at Immediate post-intervention
  Current pain intensity will be measured by a 10-cm line
The Visual Analog Scale (VAS) | Change from Baseline in Visual Analog Scale at 2 days
  Current pain intensity will be measured by a 10-cm line
Western Ontario and McMaster Universities (WOMAC) Index | Change from Baseline in WOMAC at 2 days
  Self-administered questionnaire presented in Likert-scale format
Self-Leeds Assessment of Neuropathic Symptoms and signs (S-LANSS) Scale | At Baseline
  A clinical-based instrument for identifying patients whose pain is dominated by neuropathic mechanisms
Pressure Pain Threshold (PPT) | Change from Baseline in PPT at Immediate post-intervention
  A digital pressure algometer will be used to quantify pain intensity in Kpa
Pressure Pain Threshold (PPT) | Change from Baseline in PPT at 2 days
  A digital pressure algometer will be used to quantify pain intensity in Kpa
Thermal Perception and Pain Thresholds | Change from Baseline in Thermal Perception and Pain Thresholds at Immediate post-intervention
  A Thermotest System will be used to determine thermal thresholds in degree centigrade
Thermal Perception and Pain Thresholds | Change from Baseline in Thermal Perception and Pain Thresholds at 2 days
  A Thermotest System will be used to determine thermal thresholds in degree centigrade
Hand-Held Dynamometer | Change from Baseline in Hand-Held Dynamometer at Immediate post-intervention
  A digital instrument will be used to examine isometric muscle strength of force development in pound
Hand-Held Dynamometer | Change from Baseline in Hand-Held Dynamometer at 2 days
  A digital instrument will be used to examine isometric muscle strength of force development for knee flexion and extension in pound
Standard Goniometer | Change from Baseline in Standard Goniometer at Immediate post-intervention
  Active range of motion for knee flexion and extension in degree
Standard Goniometer | Change from Baseline in Standard Goniometer at 2 days
  Active range of motion for knee flexion and extension in degree
Three-meter Timed "Up and Go" | Change from Baseline in Three-meter Timed "Up and Go" at Immediate post-intervention
  A walk test will be used to test a basic functional mobility
Three-meter Timed "Up and Go" | Change from Baseline in Three-meter Timed "Up and Go" at 2 days
  A walk test will be used to test a basic functional mobility

CONTACTS AND LOCATIONS:
Overall Officials: Ali M Alshami, Ph.D, Study Director — Imam Abdulrahman Bin Faisal University

REFERENCES:
- [Background] Creamer P, Hochberg MC. Osteoarthritis. Lancet. 1997 Aug 16;350(9076):503-8. doi: 10.1016/S0140-6736(97)07226-7. No abstract available. PMID 9274595
- [Background] Kidd BL. Osteoarthritis and joint pain. Pain. 2006 Jul;123(1-2):6-9. doi: 10.1016/j.pain.2006.04.009. Epub 2006 May 22. No abstract available. PMID 16714085
- [Background] Alghamdi MA, Olney S, Costigan P. Exercise treatment for osteoarthritis disability. Ann Saudi Med. 2004 Sep-Oct;24(5):326-31. doi: 10.5144/0256-4947.2004.326. PMID 15573841
- [Background] Gwilym SE, Pollard TC, Carr AJ. Understanding pain in osteoarthritis. J Bone Joint Surg Br. 2008 Mar;90(3):280-7. doi: 10.1302/0301-620X.90B3.20167. PMID 18310746
- [Background] Gross KD, Hillstrom H. Knee osteoarthritis: primary care using noninvasive devices and biomechanical principles. Med Clin North Am. 2009 Jan;93(1):179-200, xii. doi: 10.1016/j.mcna.2008.09.007. PMID 19059028
- [Result] Felson DT, Naimark A, Anderson J, Kazis L, Castelli W, Meenan RF. The prevalence of knee osteoarthritis in the elderly. The Framingham Osteoarthritis Study. Arthritis Rheum. 1987 Aug;30(8):914-8. doi: 10.1002/art.1780300811. PMID 3632732
- [Result] Jordan JM, Helmick CG, Renner JB, Luta G, Dragomir AD, Woodard J, Fang F, Schwartz TA, Abbate LM, Callahan LF, Kalsbeek WD, Hochberg MC. Prevalence of knee symptoms and radiographic and symptomatic knee osteoarthritis in African Americans and Caucasians: the Johnston County Osteoarthritis Project. J Rheumatol. 2007 Jan;34(1):172-80. PMID 17216685
- [Result] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497
- [Result] Oliveria SA, Felson DT, Reed JI, Cirillo PA, Walker AM. Incidence of symptomatic hand, hip, and knee osteoarthritis among patients in a health maintenance organization. Arthritis Rheum. 1995 Aug;38(8):1134-41. doi: 10.1002/art.1780380817. PMID 7639811
- [Result] Al-Arfaj A, Al-Boukai AA. Prevalence of radiographic knee osteoarthritis in Saudi Arabia. Clin Rheumatol. 2002 May;21(2):142-5. doi: 10.1007/s10067-002-8273-8. PMID 12086165
- [Derived] Alkhawajah HA, Alshami AM. The effect of mobilization with movement on pain and function in patients with knee osteoarthritis: a randomized double-blind controlled trial. BMC Musculoskelet Disord. 2019 Oct 18;20(1):452. doi: 10.1186/s12891-019-2841-4. PMID 31627723